CLINICAL TRIAL: NCT00062452
Title: Esophageal Motility and Airway Defenses Among Infants
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EMADAI (completed); R03DK061502 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2010-01

CONDITIONS: Infant, Premature, Diseases; Congenital Abnormalities; Perinatal Asphyxia
Keywords: Esophageal; Airway
MeSH Terms: conditions — Infant, Premature, Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A-1,2,3: The cohort (A) comprised of high risk infants. There were 3 sub groups studied within this cohort: (1) premature infants, (2) Infants with congenital gut anomalies, and (3) perinatal asphyxia.

SUMMARY:
Feeding difficulties and airway related consequences contribute significantly to the infant mortality and morbidity. Some of these problems may be dependent on neural control and muscular function. Prematurity, congenital anomalies and perinatal depression represent three important conditions in infants, that may have feeding and airway difficulties.Development of motility of the foregut and the adaptation during normal and disease in developing infants is unclear.

DETAILED DESCRIPTION:
With the aid of small clinical research funding from the NIDDK, in this proposal, we have developed methods to safely evaluate foregut motility in relation to breathing among high risk infants. We are using simultaneous esophageal motility studies, swallowing and respiratory measurements in this evaluation.

ELIGIBILITY:
Inclusion Criteria:

Prematurely born infants, Infants with congenital foregut anomalies, Infants with perinatal asphyxia, Ability to maintain vital signs at study,

Exclusion Criteria:

No contraindication to enteral feeding

Ages: 2 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants congenital foregut anomalies Perinatal asphyxia
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2002-05; Primary Completion 2005-04 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan R Jadcherla, MD, Principal Investigator — Nationwide Children's Hospital/The Ohio State University College of Medicine
Locations (1):
- Columbus Childrens Hospital, Columbus, Ohio, United States

REFERENCES:
- [Result] Jadcherla SR, Duong HQ, Hoffmann RG, Shaker R. Esophageal body and upper esophageal sphincter motor responses to esophageal provocation during maturation in preterm newborns. J Pediatr. 2003 Jul;143(1):31-8. doi: 10.1016/S0022-3476(03)00242-7. PMID 12915821
- [Result] Jadcherla SR, Hoffmann RG, Shaker R. Effect of maturation of the magnitude of mechanosensitive and chemosensitive reflexes in the premature human esophagus. J Pediatr. 2006 Jul;149(1):77-82. doi: 10.1016/j.jpeds.2006.02.041. PMID 16860132
- [Result] Jadcherla SR, Gupta A, Stoner E, Coley BD, Wiet GJ, Shaker R. Correlation of glottal closure using concurrent ultrasonography and nasolaryngoscopy in children: a novel approach to evaluate glottal status. Dysphagia. 2006 Jan;21(1):75-81. doi: 10.1007/s00455-005-9002-7. PMID 16786412
- [Result] Jadcherla SR. Manometric evaluation of esophageal-protective reflexes in infants and children. Am J Med. 2003 Aug 18;115 Suppl 3A:157S-160S. doi: 10.1016/s0002-9343(03)00215-8. PMID 12928093
- [Result] Jadcherla SR, Duong HQ, Hofmann C, Hoffmann R, Shaker R. Characteristics of upper oesophageal sphincter and oesophageal body during maturation in healthy human neonates compared with adults. Neurogastroenterol Motil. 2005 Oct;17(5):663-70. doi: 10.1111/j.1365-2982.2005.00706.x. PMID 16185304
- [Result] Gupta A, Jadcherla SR. The relationship between somatic growth and in vivo esophageal segmental and sphincteric growth in human neonates. J Pediatr Gastroenterol Nutr. 2006 Jul;43(1):35-41. doi: 10.1097/01.mpg.0000226368.24332.50. PMID 16819375